CLINICAL TRIAL: NCT06696716
Title: ONO-4059-10:Multicenter, Placebo-controlled, Randomized, Double-blind, Phase 3 Study in Patients With Steroid-resistant Pemphigus (BRILLIANT Study)
Brief Title: ONO-4059 Study in Patients With Steroid-resistant Pemphigus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4059-10; jRCT2031220043 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-11-07; First posted 2024-11-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pemphigus; Steroid-resistant Pemphigus
MeSH Terms: conditions — Pemphigus | interventions — tirabrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-4059 (Active Comparator)
  Interventions: Drug: ONO-4059
- Placebo (Placebo Comparator)
  Interventions: Drug: ONO-4059 placebo

INTERVENTIONS:
Drug: ONO-4059 — Tirabrutinib is a Bruton's Tyrosine Kinase Inhibitor. Tirabrutinib will be administered orally at a dose of 80 mg once daily after a meal (breakfast, lunch, or dinner).
  Other Names: Tirabrutinib hydrochloride
  Arms: ONO-4059
Drug: ONO-4059 placebo — Placebo will be administered orally once daily after a meal (breakfast, lunch, or dinner).
  Arms: Placebo

SUMMARY:
ONO-4059-10:Multicenter, placebo-controlled, randomized, double-blind, Phase 3 study in patients with steroid-resistant pemphigus

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pemphigus
* Patients with a re-increase in the pemphigus disease area index (PDAI) score before oral corticosteroid tapering to 10mg/day of prednisolone (PSL) equivalent

Exclusion Criteria:

* Patients with an active infection
* Patients with malignancy
* Patients with past history of serious allergy or anaphylaxis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a Complete response (CR) or Partial response (PR) at 52 weeks, and maintaining complete/partial remission at 52 weeks from initial remission achievement. | 52 weeks
  CR: Absence of pemphigus-related blisters or new erythema that lasts for 8 weeks during treatment with ONO-4059 plus an oral corticosteroid (≤10 mg/day prednisolone-equivalent) or minimal adjunctive therapy.
  PR: Occurrence of only a transient lesion that resolves within 1 week without an increased dose of an oral corticosteroids, without treatment, or with a topical corticosteroid, etc., during treatment with ONO-4059 plus an oral corticosteroid (≤10 mg/day prednisolone-equivalent) or minimal adjunctive therapy for 8 weeks.

SECONDARY OUTCOMES:
Remission rate | 52 weeks
  remission rate [proportion of subjects who achieve complete or partial remission], complete remission rate, partial remission rate
Pemphigus Disease Area Index (PDAI) score | 52 weeks
  Pemphigus Disease Area Index (PDAI). PDAI activity score cutoffs were defined as 0 to 8 for mild, 9 to 24 for moderate, and 25 or higher for severe disease.
Efficacy 1 rate (proportion of subjects for whom the definition of efficacy 1 is applicable) | 52 weeks
  Definition of efficacy 1: Decreases in PDAI score and oral corticosteroid dose from baseline
Efficacy 2 rate (proportion of subjects for whom the definition of efficacy 2 is applicable) | 52 weeks
  Definition of efficacy 2: PDAI score is 0 and oral corticosteroid dose <= 10 mg/day
Disease control rate (proportion of subjects for whom the definition of disease control is applicable) | 52 weeks
  Definition of disease control: Formation of nascent lesions stops and existing lesions begin to resolve
Rescue therapy rate | 52 weeks
  Proportion of subjects who received rescue therapy
Pemphigus autoantibody titer | 52 weeks
  Anti-desmoglein 1 antibodies, anti-desmoglein 3 antibodies
Oral corticosteroid dose | 52 weeks
  At the equivalent dose of prednisolone
QOL evaluation | 52 weeks
  The Dermatology Life Quality Index (DLQI) score is measured by questionnaire.
Adverse events and adverse drug reactions | 52 weeks
Clinical laboratory tests | 52 weeks
  Number of participants with clinical laboratory abnormalities (including haematology, clinical chemistry and urinalysis).
12-lead ECG | 52 weeks
  Heart rate, RR interval, PR interval, QRS duration, QT interval and QTcF
Vital signs | 52 weeks
  Systolic/diastolic blood pressure
Vital signs | 52 weeks
  Body temperature
Immunological tests | 52 weeks
  Immunoglobulin G and its subclasses (IgG 1, 2, 3, and 4), immunoglobulin M, immunoglobulin A, peripheral blood B-cell count, and peripheral blood T-cell count
Plasma ONO-4059 concentration | 52 weeks
Immunophenotyping | 52 weeks
  Level of naive-B cell, memory-B cell, plasmablast etc.
Cytokines and chemokines | 52 weeks
  Level of tumor necrosis factor-α, interleukin (IL)-8, IL-13, IL-17, C-X-C motif chemokine ligand 13 etc.
RNA sequencing | 52 weeks
Anti-virus antibody | 52 weeks
Recurrence rate (the proportion of subjects meeting the definition of recurrence) and time to recurrence | 52 weeks
  Definition of recurrence: In patients with controlled disease, the presence of three or more new lesions in a month that do not spontaneously resolve within a week, or the expansion of existing lesions Definition of time to recurrence: The period from achieving disease control to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (25):
- Japan (25):
  - Ichinomiya Municipal Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Ehime University Hospital, Ehime
  - Kurume University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gunma University Hospital, Gunma
  - Hokkaido University Hospital, Hokkaido
  - Kagoshima University Hospital, Kagoshima
  - St.Marianna University School of Medicine Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Yokohama City University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Kawasaki Medical School Hospital, Okayama
  - University of the Ryukyus Hospital, Okinawa
  - Kindai university hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Saitama Medical Center, Saitama
  - Shiga University of Medical Science Hospital, Shiga
  - Jichi Medical University Hospital, Tochigi
  - Keio University Hospital, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Tokyo Women'ｓ Medical University Hospital, Tokyo
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No